CLINICAL TRIAL: NCT06998823
Title: The Effect of Survival, Response and Microbiota Change in Different Therapy Under Probiotic Supplement (Clostridium Butyricum) in Patient With Malignant Tumor
Brief Title: The Effect of Survival, Response and Microbiota Change in Different Therapy Under Probiotic Supplement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, ChengHaoTsai, Professor Attending Physicians, Chang Gung Memorial Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 202201539A3
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Probiotics; Cancer, Therapy-Related
Keywords: Probiotics; Immunotherapy; Targeted Therapy; Chemotherapy
MeSH Terms: conditions — Neoplasms, Second Primary | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: 90 participants will intake 90days Probiotics (Clostridium butyricum). Investigators also collect these participants' stool for intestinal microbiota, do the liver fibrosis evaluting and blood drawing for the phenoage assessment before taking probiotics, when there are changes in condition during treatment, and after probiotics.
  30 participants don't intake Probiotics. Investigators also collect these patients twice stool for intestinal microbiota, do the fibroscan evaluting and blood drawing for the pheniage assessment before and after Probiotics: 1st time (before cancer treatment), 2nd time (when there are changes in condition during treatment) and 3rd time (after 90days cancer treatment later).
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): Participants don't intake Probiotics (Clostridium butyricum). Investigators also collect these patients twice stool for intestinal microbiota, do the fibroscan evaluting and blood drawing for the pheniage assessment before and after Probiotics: 1st time (before cancer treatment), 2nd time (when there are changes in condition during treatment) and 3rd time (after 90days cancer treatment later).
- experimental (Experimental): Participants will intake 90days Probiotics (Clostridium butyricum). Investigators also collect these patients' stool for intestinal microbiota, do the liver fibrosis evaluting and blood drawing for the phenoage assessment before taking probiotics, when there are changes in condition during treatment, and after probiotics
  Interventions: Combination Product: Probiotics

INTERVENTIONS:
Combination Product: Probiotics — Participants will intake 90days Probiotics
  Arms: experimental

SUMMARY:
Probiotics are a group of viable microorganisms including bacteria and yeasts that if consumed in sufficient amounts, may afford health benefits to the host. The major advantage of probiotic administration is its ability to maintain gut microbial homeostasis, reduce pathogenic microorganisms in the GI tract, and restores homeostasis of intestinal microorganisms. Moreover, by modulating microbiota and immune responses, decreasing bacterial translocation, promoting the function of the gut barrier, inducing anti- inflammatory properties, triggering anti-pathogenic activity, and decreasing tumor development and metastasis, probiotics might contribute to the prevention and treatment of GI cancers and lung cancer. Considering the potential roles of Helicobacter pylori (H. pylori) in the initiation of colorectal and gastric cancers, the possible properties of probiotics against GI neoplasm in humans have been investigated in relation to their suppressive effects on H. pylori. The gut microbiota also has proved to in the response and resistance to immunotherapy. By triggering immune activity, probiotics, as functional dietary supplements, may mitigate neoplastic predisposition and development of GI cancers. Clostridium butyricum is a spore-forming bacillus named for its capacity to produce high amounts of butyric acid and is found in soil. Clostridium butyricum MIYAIRI 588 strain (MIYA-BM) is widely used as probiotic therapy to improve symptoms related to dysbiosis such as constipation, nonantimicrobial diarrhea, and anti- microbial-associated diarrhea in Japan and China. Clostridium butyricum increases beneficial bacteria, especially lactobacilli and bifidobacteria. Bifidobacterium promotes antitumor immunity and facilitates efficacy of antitumor treatment. The antitumor treatments are differed to three types: immune checkpoint blockade, target therapy and chemotherapy. Thus, investigators hypothesized that probiotic Clostridium butyricum therapy (CBT) may enhance the therapeutic efficacy of anti-tumor therapy through the modulation of gut microbiota. Investigators will discuss the different kinds of anti-tumor effect in survival and response after probiotic supplement.

DETAILED DESCRIPTION:
Probiotics are a group of viable microorganisms including bacteria and yeasts that if consumed in sufficient amounts, may afford health benefits to the host. The major advantage of probiotic administration is its ability to maintain gut microbial homeostasis, reduce pathogenic microorganisms in the GI tract, and restores homeostasis of intestinal microorganisms. Moreover, by modulating microbiota and immune responses, decreasing bacterial translocation, promoting the function of the gut barrier, inducing anti- inflammatory properties, triggering anti-pathogenic activity, and decreasing tumor development and metastasis, probiotics might contribute to the prevention and treatment of GI cancers and lung cancer. Considering the potential roles of Helicobacter pylori (H. pylori) in the initiation of colorecta and gastric cancers, the possible properties of probiotics against GI neoplasm in humans have been investigated in relation to their suppressive effects on H. pylori. The gut microbiota also has proved to in the response and resistance to immunotherapy. By triggering immune activity, probiotics, as functional dietary supplements, may mitigate neoplastic predisposition and development of GI cancers.

Clostridium butyricum is a spore-forming bacillus named for its capacity to produce high amounts of butyric acid and is found in soil. Clostridium butyricum MIYAIRI 588 strain (MIYA-BM) is widely used as probiotic therapy to improve symptoms related to dysbiosis such as constipation, nonantimicrobial diarrhea, and anti- microbial-associated diarrhea in Japan and China. Clostridium butyricum increases beneficial bacteria, especially lactobacilli and bifidobacteria. Bifidobacterium promotes antitumor immunity and facilitates efficacy of antitumor treatment. The antitumor treatments are differed to three types: immune checkpoint blockade, target therapy and chemotherapy. Thus, investigators hypothesized that probiotic Clostridium butyricum therapy (CBT) may enhance the therapeutic efficacy of anti-tumor therapy through the modulation of gut microbiota. Investigators will discuss the different kinds of anti-tumor effect in survival and response after probiotic supplement.

This is a prospective study. Investigators evaluate 120 participants with advanced malignant tumor consecutively treated with anti-tumor therapy in routine clinical practice at New Taipei Municipal Tucheng Hospital and Linkou branch of Chang Gung Memorial Hospital. These 120 participants were equal to separate three groups: immune therapy, target therapy and chemotherapy. Each group will have 30 participants receiving Probiotics and 10 participants without Probiotics. The include criteria is participants agree to probiotics used. The exclude criteria ia participants refuse probiotics used.90 participants will intake 90days Probiotics (Clostridium butyricum). Investigators also collect these participants' stool for intestinal microbiota, do the liver fibrosis evaluting and blood drawing for the phenoage assessment before taking probiotics, when there are changes in condition during treatment, and after probiotics .

ELIGIBILITY:
Inclusion Criteria:

1. age≧20
2. participants with cancer therapy and agree to sign informed consent
3. Cancer confirmed by clinical or pathological diagnosis

Exclusion Criteria:

1. age<20
2. Pregnant or breastfeeding women

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2025-10-25 (Estimated); Study Completion 2026-11-08 (Estimated)

PRIMARY OUTCOMES:
phenoage score | baseline
  collect 10 mL of peripheral blood, and caculate the phenoage
phenoage score | 3 month
  collect 10 mL of peripheral blood, and caculate the phenoage
Metagenomic shotgun sequencing | baseline
  Collect stool samples to analyze the types and unique characteristics of microorganisms
Metagenomic shotgun sequencing | 3 month
  Collect stool samples to analyze the types and unique characteristics of microorganisms
Liver Fibrosis score | baseline
  do the liver fibrosis assessment by using fibroscan for evaluating the impact on liver fibrosis after taking Probiotics and caner therapy.
Liver Fibrosis score | 3 month
  do the liver fibrosis assessment by using fibroscan for evaluating the impact on liver fibrosis after taking Probiotics and caner therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Hsun Hsieh, PhD, Principal Investigator — Division of Oncology, Chang Gung Memorial Hospital
Locations (1):
- New Taipei City TuCheng Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No